CLINICAL TRIAL: NCT02627326
Title: Evaluation of Effectiveness of Chlorhexidine Intracanal Medicament on Periodontal Healing in Concomitant Endodontic and Periodontal Disease With Communication : A Randomized Controlled Clinical Trial
Brief Title: Chlorhexidine Intracanal Medicament in Periodontal Healing in Concomitant Endo Perio Lesion With Communication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: perio1
Record Dates: First submitted 2015-12-06; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Periodontal Pocket; Tooth,Non Vital
Keywords: chlorhexidine; endodontic treatment
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Interventions done in 30 patients and included conventional endodontic treatment (ET) and periodontal surgery . After 3 months of completion of endodontic therapy without using 2%chlorhexidine gluconate gel intracanal medicament , periodontal surgery in the form of open flap debridement (OFD) was performed.
  Interventions: Procedure: open flap debridement
- Group 2 Chlorhexidine (Active Comparator): Interventions done in 30 patients and included intracanal medicament . After biomechanical preparation of root canal, 2%Chlorhexidine gluconate gel as an intracanal medicament was placed in root canal from pulp chamber to apex for 3 months (replacing every month). After 3 months,periodontal surgery in the form of open flap debridement (OFD) was performed in the respective tooth and medicament was changed and placed further for 3 months (replacing every month). Obturation was done after 3 months of OFD.
  Interventions: Procedure: open flap debridement

INTERVENTIONS:
Procedure: open flap debridement — periodontal surgery in the form of open flap debridement was done in both the groups
  Other Names: OFD

SUMMARY:
The aim of this prospective randomized controlled clinical trial is to evaluate the effectiveness of chlorhexidine intracanal medicament along with periodontal treatment in concomitant endodontic periodontal lesions with communication in terms of periodontal healing. Forty-seven patients were randomly divided into: group 1: conventional endodontic treatment with open flap debridement (OFD after 3 month of endodontic treatment) were performed, in group 2: endodontic treatment with 2% chlorhexidine gel (CHX) as an intracanal medicament placed in root canals and after 3 month OFD were performed. Primary outcome variables included probing pocket depth, clinical attachment level and bleeding on probing.

DETAILED DESCRIPTION:
INTRODUCTION:

Treatment decision-making and prognosis of endodontic-periodontal lesion is primarily dependent on the diagnosis of the specific endodontic or periodontal disease. Although the treatment of endodontic and periodontal lesions arouse a lot of confusions and speculations. Wherein, endodontic-periodontal combined lesion is a clinical dilemma because making a differential diagnosis and deciding a prognosis are difficult. Also, the success of such lesions depends on the elimination of both of these disease processes as the endodontic therapy results in healing of the endodontic component of involvement while the prognosis of tooth would finally depend on the healing of the periodontal structures.

Interventional studies also reported negative influence on the periodontal healing in presence of infected root canal system, after providing periodontal treatment. However, in addition to this, the outcome of endodontic treatment may be affected if the root canal filling is placed while there is still a periodontal infection present that communicates with the root canal system since cross-seeding through the apical or lateral foramina is possible. Despite thorough cleaning and disinfection of the root canal system during endodontic treatment, bacteria from the periodontal lesion may re-invade the root canal system since root canal fillings do not seal canals completely.

The elimination of microorganisms from infected root canal is a complicated task involving the use of various instrumentation techniques, irrigation regimens and intracanal medicaments. Gomes et al observed that 2% chlorhexidine (CHX) showed maximum zone of inhibition against porphyromonas gingivalis, enterococcus faecalis, actinomyces viscosus and candida albicans followed by a combination of calcium hydroxide and CHX, and least with calcium hydroxide alone. A clinical study carried out by zamany et al showed that 2% CHX solution used as a final irrigant, significantly decreased bacterial loads in root canal. Additional advantages of chlorhexidine are its retentive character in root canal dentin and its relatively low toxicity and its effect on periodontal healing has been well known. Based on these observations, it may be hypothesized that intracanal medicament may act as a controlled released drug which could be used as an adjunct to periodontal surgical therapy .

Thus the present study was conducted to evaluate the effectiveness of chlorhexidine intracanal medicament along with periodontal surgical therapy on periodontal healing in concomitant endodontic and periodontic disease with communication.

MATERIAL AND METHODS:

This study was conducted in Department of Periodontics and Oral Implantology in collaboration with Department of Conservative Dentistry and Endodontics, Post Graduate Institute of dental sciences (PGIDS), Rohtak.

The study protocol was carried out in accordance with the ethical standards outlined in the Helsinki declaration 1964, as revised in 2013.39. The protocol was approved by the Institutional Review Board, Pt. B. D. Sharma University of Health Sciences, Rohtak and the ethical approval (IEC/2014/115) was obtained from the ethical committee of PGIDS, Rohtak.

STUDY POPULATION:

This study was designed as a prospective randomized double blind controlled clinical trial. Patients were recruited from regular outpatient department of the periodontics, endodontics and oral diagnosis, PGIDS, Rohtak. A total of 250 patients were examined and out of them 47 patients suffering from chronic periodontitis having combined endodontic periodontal lesion with communication and meeting the inclusion criteria were treated from May 2014 to September 2015.

INCLUSION CRITERIA

Patients of age between 18-55 years with generalized chronic periodontitis and having at least one tooth with concomitant endodontic periodontal lesion with communication including following features:

* a clinical and radiographic diagnosis of concomitant endodontic periodontal lesion
* Wide base pocket, deep probing pocket depth
* Non vital tooth with periapical radiolucency
* Radiographic alveolar bone (marginal bone) destruction with apical communication EXCLUSION CRITERIA- Systemic illness known to affect the periodontium or outcome of periodontal therapy.
* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy or bisphosphonates.
* Patients allergic to medication (local anaesthetic, antibiotics, NSAID).
* Patients with acute symptoms.
* Pregnant or lactating females.
* Smokers (current and past) and tobacco chewers.
* Grade 3 mobile teeth.
* Unrestorable tooth.
* Root resorption.
* Fractured/perforated roots.
* Developing permanent tooth.
* Abutments.
* Previously root canal filled.
* Patients with aggressive periodontitis
* History of periodontal treatment within 6 months prior to study. After confirming the eligibility, written and verbal informed consent was obtained from each patient.

METHODOLOGY:

Patients were randomly allocated to one of the two treatment groups according to a computer-generated randomization list. It was ensured that neither the investigator nor the patient was aware of the treatment protocol at the time of patient allocation. From each patient only one tooth was selected.

Group 1 (n = 23 teeth/23 patients), endodontic treatment (ET) and full mouth scaling and root planing (SRP) were performed simultaneously. After 3 months of commencement of endodontic therapy, periodontal surgical treatment in the form of open flap debridement (OFD) was performed.

Group 2 (n = 24 teeth/24 patients), endodontic treatment (ET) and full mouth scaling and root planing (SRP) were started simultaneously. After biomechanical preparation of root canal, CHX intracanal medicament was placed in root canal from pulp chamber to apex for 3 months (replacing every month). After 3 months, open flap debridement (OFD) was performed in the respective tooth and medicament was changed and placed further for 3 months (replacing every month). Obturation was done after 3 months of OFD.

Clinical Data Collection: Endodontic evaluation - Pulp sensibility testing was performed with a combination of heat test (heated gutta-percha), cold test (Endo-Frost, Coltene, Whaledent) and electric pulp test (Digitest D626D, Parkell electronics, New York). Teeth not responding to both thermal and electric test were considered non vital.

Radiographic evaluation - Radiographs with paralleling cone technique were taken with standardized exposure parameters (70kvp, 3.5mAs, and 0.2 seconds) by single operator using dental x-ray machine .

PERIODONTAL EXAMINATION

CLINICAL PARAMETERS:

Full mouth indices recorded at baseline Plaque index (Silness and Loe) (PI) Gingival index (Loe and Silness) (GI) Bleeding on probing (BOP) Probing pocket depth (PPD) Clinical attachment level (CAL) Site specific ( endo- perio involved tooth) indices Plaque index

* Gingival index
* Relative Probing pocket depth
* Relative clinical attachment loss
* Bleeding on probing
* Tooth mobility
* Relative gingival marginal level Clinical parameters were recorded at baseline, 3 months, 6 months and 9 months. Each of the tooth was assessed at four sites (mesiobuccal, midbuccal, distobuccal, midlingual) for PI and GI and six sites (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual) for PPD, CAL, BOP during full mouth complete periodontal examination.

PERIODONTAL NON SURGICAL PROCEDURE: All the patients enrolled for the study at the initial visits undergo non surgical periodontal treatment in the form of scaling and root planing (SRP) which was performed with ultrasonic scaler and hand instruments. SRP was completed in two to three sessions along with education and motivation to maintain the health of periodontium.

CONVENTIONAL ENDODONTIC PROCEDURE: Simultaneously along with non surgical periodontal treatment, root canal treatment was performed by experienced endodontist using a standardized protocol. The standard procedures for all cases included local anaesthesia (2% lidocaine with 1:80,000 epinephrine), rubber dam isolation, pulp extirpation and standard access cavity preparation. After flooding the pulp chamber with 3% sodium hypochlorite (NaOCl; Sainsbury plc, London, UK), canal negotiation & apical patency was achieved with #10 or #15K-files. Coronal flare was created with # 2 and #3 Gates-Glidden drills (Dentsply Maillefer, Tulsa, OK). Working length of each canal was established with Root-ZX apex locator (J Morita, Irwine, CA) and verified with radiographs. Canal instrumentation was performed with K files in a crown-down technique. The master apical file size was set at 3 sizes larger than the first binding file at working length. Instrumentation was carried out in conjunction with copious irrigation with 3% sodium hypochlorite using 27 gauge needles.

In group 1, lentulospiral was used to fill all canals with calcium hydroxide and tooth was sealed with Intermediate Restorative Material and patients were scheduled for a second appointment to obdurate the root canals within 10 days. At the next appointment, calcium hydroxide paste was removed by using circumferential filing with Hedstrom-type files and copious irrigation with 3% sodium hypochlorite followed by 5.0 mL 17% ethylenediaminetetraacetic acid and a final rinse of 5.0 mL of 3% sodium hypochlorite. The canals were dried with sterile paper points and obturated by using lateral condensation technique with gutta-percha and zinc oxide sealer and permanent filling was placed in form of silver amalgam.

In group 2, 2% CHX gel was placed and filled in the root canal space up to apex using 27 gauge endodontic syringe after cleaning with 17% EDTA and saline and tooth was coronally sealed with glass inomer cement (Version 2, Shofu, Kyoto, Japan). This intracanal medicament was changed every 1 month for 6 months and after 6 months canals were obturated same as in group 1.

PERIODONTAL SURGICAL PROCEDURE: 5% povidone iodine solution was used for extraoral antisepsis and intraoral antisepsis. After achieving local anaesthesia (2% lidocaine with 1:80,000 epinephrine), buccal and lingual/palatal intracrevicular incision were made with BP blade number 15 and full thickness mucoperiosteal flaps were reflected including neighbouring teeth. Meticulous defect debridement and root planing was carried out using area specific gracey curettes and scalers to remove all the granulation tissue and deposits. After instrumentation, the root surface was washed with saline solution in attempt to remove any remaining detached fragments from the defect and surgical field. After debridement mucoperiosteal flaps was repositioned and secured by using 3-0 non absorbable black silk surgical suture. The surgical area was protected and covered with non eugenol periodontal dressing (coe pak, GC America Inc, USA) and post operative instructions were given.

FOLLOW UP: All parameters were re-evaluated and recorded at baseline, 3 month, 6 month and 9 month of follow up.

STATISTICAL ANALYSES: Data were found to be non-normally distributed. Intragroup differences were analysed by Wilcoxan Signed Rank test. Intergroup comparison of measurements were analysed by Mann-Whitney U test..

Partial correlation analysis was done to analyse the correlation between the type of treatment provided and clinical variables (at the 9 months of follow up) after controlling of potential confounders PI and age. All the variables that had shown a significant correlation were included in logistic regression analysis. Models were adjusted for the co-variates. The Hosmer-Lemeshow statistic was applied to verify the diagnosis of the goodness-of-fit regression model employed. All statistical analyses were two tailed with significance level at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age between 18-55 years with generalized chronic periodontitis and having at least one tooth with concomitant endodontic periodontal lesion with communication including following features:

  * a clinical and radiographic diagnosis of concomitant endodontic periodontal lesion
  * Wide base pocket, deep probing pocket depth
  * Non vital tooth with periapical radiolucency
  * Radiographic alveolar bone (marginal bone) destruction with apical communication Criteria for generalized chronic periodontitis [≥30% sites involved with clinical attachment loss (CAL) 1-2mm (mild) or 3-4mm (moderate) or ≥5mm (severe)]40 Patient should have more than 20 teeth

Exclusion Criteria:Systemic illness known to affect the periodontium or outcome of periodontal therapy.

* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy or bisphosphonates.
* Patients allergic to medication (local anaesthetic, antibiotics, NSAID).
* Patients with acute symptoms.
* Pregnant or lactating females.
* Smokers (current and past) and tobacco chewers.
* Grade 3 mobile teeth.
* Unrestorable tooth.
* Root resorption.
* Fractured/perforated roots.
* Developing permanent tooth.
* Abutments.
* Previously root canal filled.
* Patients with aggressive periodontitis
* History of periodontal treatment within 6 months prior to study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
probing pocket depth | 9 months
clinical attachment level | 9 months
bleeding on probing | 9 months